CLINICAL TRIAL: NCT01967251
Title: A Randomized, Triple Blind, Placebo-controlled, Parallel-group Trial to Assess the Efficacy, Safety and Dose Response of Udenafil for 12 Weeks in Mexican Patients With Benign Prostatic Hyperplasia and Erectile Dysfunction
Brief Title: Efficacy, Safety and Dose-response of Udenafil in Patients With Benign Prostatic Hyperplasia and Erectile Dysfunction
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MX030; U1111-1146-1278 (Other: World Health Organization)
Record Dates: First submitted 2013-10-17; First posted 2013-10-22 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Erectile Dysfunction; Benign Prostatic Hyperplasia
Keywords: Prostatic Hyperplasia; Phosphodiesterase 5 inhibitors; Erectile DysfunctionDrug Therapy
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Hyperplasia | interventions — udenafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Udenafil 25 mg (Experimental): Udenafil 25 mg, tablets, orally, once daily for 12 weeks.
  Interventions: Drug: Udenafil
- Udenafil 50 mg (Experimental): Udenafil 50 mg, tablets, orally, once daily for 12 weeks.
  Interventions: Drug: Udenafil
- Udenafil 75 mg (Experimental): Udenafil 75 mg, tablets, orally, once daily for 12 weeks.
  Interventions: Drug: Udenafil
- Placebo (Placebo Comparator): Udenafil placebo-matching tablets, orally, once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Udenafil — Udenafil tablets
  Arms: Udenafil 25 mg; Udenafil 50 mg; Udenafil 75 mg
Drug: Placebo — Udenafil placebo-matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, dose-response and safety of udenafil 25 mg, 50 mg and 75 mg every day (q.d.) for 12 weeks in the treatment of lower urinary tract symptoms (LUTS) associated with benign prostatic hyperplasia (BPH and for the treatment of erectile dysfunction (ED).

DETAILED DESCRIPTION:
The drug being tested in this study is called Udenafil. Udenafil is being tested to treat lower urinary tract symptoms (LUTS) associated with benign prostatic hyperplasia (BPH) and for the treatment of erectile dysfunction (ED). This study will look at the change in lower urinary tract symptoms (LUTS) associated with benign prostatic hyperplasia (BPH) and in erectile dysfunction (ED) in people who take Udenafil.

The study will enroll approximately 950 patients. Participants taking BPH or ED medication will enter a 4-week wash out period. Patients not previously treated and those who accomplished the wash out period will enter a placebo (dummy inactive pill) lead-in period of another 4 weeks. Participants will then be randomly assigned (by chance, like flipping a coin) to one of the four treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Udenafil 25 mg
* Udenafil 50 mg
* Udenafil 75 mg
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient

All participants will be asked to take one tablet at the same time each day throughout the study, and will be asked to keep a Sexual Encounter Profile (SEP) diary.

This multi-centre trial will be conducted in Mexico. The overall time to participate in this study is up to 20 weeks. Participants will make 6 visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Men ≥ 45 years of age.
2. Sexually active, with a stable female partner with whom the participant expects to have a relationship for the entire duration of the study.
3. The participant has benign prostatic hyperplasia with lower urinary tract symptoms (BPH-LUTS) according to clinical diagnostic criteria, with ≥ 6 months of evolution at the screening visit.
4. Clinical history of erectile dysfunction (ED) (defined as the inability to achieve or maintain the penile erection to achieve a satisfactory sexual relationship) of at least 3 months of evolution.
5. Freely given informed consent at the screening visit (an essential requirement to participate in the study).
6. Bladder obstruction defined by maximal flow rate (Qmax) of 4-15 mI/sec (with a premicturition volume of 150 to 550 mL evaluated by ultrasound, with a minimum micturition volume of 125 mL) at Visit I immediately prior to active treatment initiation.
7. Total score of ≥ 13 points in the InternationaI Prostate Symptom Score (IPSS) questionnaire at Visit 1, immediately prior to active treatment initiation.

Exclusion Criteria:

1. Participants that are currently taking nitrates, antiandrogens, estrogens, luteninizing hormone-releasing hormone agonist/antagonist, or anabolic steroids at study entry. Participants that are taking a stable dose level of testosterone are not excluded.
2. Post-void residual (PVR) volume ≥ 300 mL, as assessed by ultrasound at the Visit 1.
3. Prostate-specific antigen (PSA) ≥ 10.0 ng/mL at the Visit 1.
4. PSA of 4.0 - 10.0 ng/ml if free PSA is < 0,25 (25%) at Visit 1.
5. Clinical evidence of prostate cancer.
6. Glycosylated hemoglobin (Hb1Ac) > 10 % at study entry.
7. Patients who have undergone bladder catheterization due to acute urine retention.
8. Medical history or clinical evidence of any pelvic, bladder or urinary tract condition, or urinary retention that, as judged by the urologist, might compromise protocol compliance.
9. Any surgical procedure in the lower urinary tract (including prostate biopsy) within 30 days prior to the Screening Visit.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Total International Prostate Symptom Score (IPSS) | Baseline to Week 12
  The IPSS is an 8 question (7 symptom questions + 1 quality of life question) tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of the disease benign prostatic hyperplasia (BPH). The 7 symptoms questions include feeling of incomplete bladder emptying, frequency, intermittency, urgency, weak stream, straining and nocturia, each referring to during the last month, and each involving assignment of a score from 1 to 5 for a total of maximum 35 points. The 8th question of quality of life is assigned a score of 1 to 6. The total score correlates as follows: 0-7 mildly symptomatic; 8-19 moderately symptomatic; 20-35 severely symptomatic.
Change from Baseline in Erectile Function Domain of the International Index of Erectile Function (IIEF) | Baseline and Week 12
  The IIEF is a standardised and validated 15-item self-evaluation scale that provides pre-post treatment clinic evaluations of erectile function, orgasmic function, sexual desire, satisfaction in sexual intercourse and general satisfaction. The Erectile Function domain (6-item) provides pre-post treatment evaluations of erectile function.

SECONDARY OUTCOMES:
Participants with Adverse Events | 12 weeks
  AEs will be evaluated by monitoring participants vital signs, laboratory tests (blood chemistry, hematology, coagulation and serology tests, urianalysis), electrocardiography (ECG).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (8):
- Mexico (8):
  - Chihuahua City, Chihuahua
  - Guadalajara, Jalisco
  - Mexico City, Mexico City
  - Morelia, Michoacán
  - Cuernavaca, Morelos
  - Monterrey, Nuevo León
  - Cholula, Puebla
  - México, State of Mexico